CLINICAL TRIAL: NCT02140619
Title: Affect of Multiple Health Education Interventions on Secondary Prevention Medication Persistence and Clinical Prognosis of Ischemic Stroke Patients: a Prospective Cohort Study
Brief Title: Affect of Multiple Health Education on Medication Persistence and Clinical Prognosis of Ischemic Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: yongjun wang (Other Government)
Collaborators: Ministry of Science and Technology of the People´s Republic of China (Other Government)
Responsible Party: Sponsor-Investigator, yongjun wang, Professor,Vice president of Beijing Tiantan Hospital, Ministry of Science and Technology of the People´s Republic of China
Organization: Ministry of Science and Technology of the People´s Republic of China (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TTYY-20131201
Record Dates: First submitted 2014-05-05; First posted 2014-05-16 (Estimated); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: Ischemic Stroke; Medication Persistence
Keywords: ischemic stroke; Medication Persistence; outcome
MeSH Terms: conditions — Ischemic Stroke; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- multiple health education interventions (Active Comparator): The group will receive health education manuals and Digital Video Disc (DVD) during hospitalization and regular text message during 1 year after discharge.
  Interventions: Behavioral: multiple health education interventions
- conventional health education (Placebo Comparator): The second group will receive conventional health education during hospitalization except health education manuals, text message and Digital Video Disc (DVD)
  Interventions: Behavioral: multiple health education interventions

INTERVENTIONS:
Behavioral: multiple health education interventions

SUMMARY:
The study aimed to demonstrate the relationship between secondary prevention medication persistence and clinical prognosis of ischemic stroke patients at 3,6,12 months

DETAILED DESCRIPTION:
The study is a prospective, multicenter, hospital-based study on secondary prevention for patients with ischemic cerebrovascular diseases between May 2014 and June 2015. Physicians from 24 hospitals in Beijing underwent a standard secondary prevention training of ischemic cerebrovascular diseases by professional training, instruction manuals, stratification management software. In order to improve the persistence of taking preventive secondary medicine, IS patients from these 24 hospitals received healthy education through manuals and Digital Video Disc about health education during hospitalization and acquired secondary preventive knowledge of ischemic cerebrovascular diseases through regular health education messages during 6 months after discharge. Patients with IS from other 6 hospitals were used as a control, and no such intervention was given to them.

Telephone follow-up was performed at 3 months, 6 months, and 1 year after the onset of cerebral infarction, during which the use of antiplatelet and statins drugs and recurrence of IS were recorded. Patients who took antiplatelet drugs or statins at three follow-ups were regarded as persistent antiplatelet drugs or statins taking within one year after the onset of the disease. The main prognostic indicator was the recurrence of IS and persistence of antiplatelet and statins medication within 1 year, and the main purpose was to explore the impact of persistent statins and antiplatelet medication use on IS recurrence.

ELIGIBILITY:
Inclusion Criteria:

1. Adult subjects (male or female ≥18 years);
2. Acute ischemic stroke occured within 14 days of symptoms onset
3. Patients signed informed consent
4. Patients have a cell phone and have the ability to receive and view messages

Exclusion Criteria:

1. Non-cerebrovascular events or hemorrhagic stroke
2. Patients have serious heart, liver, kidney dysfunction or coagulation disorders
3. Patients have circumstances that may affect the follow-up such as disturbance of consciousness, severe depression or other mental disorders, aphasia
4. Modified Rankin Scale score at discharge ≥3
5. Those who are participating in other clinical trials
6. Those who can not guarantee with the completion of 1 year follow-up after enrollment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3111 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2015-06-28 (Actual); Study Completion 2015-09-30 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who continued taking antiplatelet drugs at three months after stroke onset, and proportion of patients who continued taking statins drugs at three months after stroke onset. | 3 months after stroke onset
  Medication persistence at 3 months. Persistence is defined as continuing a therapy or class of therapy from discharge to the 3 months follow-up. Subjects prescribed an individual medication at discharge but who were not taking that medication at follow up were defined as "nonpersistent". Persistence for the specified medication classes (antiplatelet, statins) was defined in the same way; however, subjects were considered persistent if there was a switch to another medication within the same class.
Proportion of patients who continued taking antiplatelet drugs at six months after stroke onset, and proportion of patients who continued taking statins drugs at six months after stroke onset. | 6 months after stroke onset
  Medication persistence at 6 months. Persistence at 6 months is defined as continuing a therapy or class of therapy at 6 months follow-up. Subjects prescribed an individual medication at discharge but who were not taking that medication at follow up were defined as "nonpersistent". Persistence for the specified medication classes (antiplatelet, statins) was defined in the same way; however, subjects were considered persistent if there was a switch to another medication within the same class.
Proportion of patients who continued taking antiplatelet drugs at 12 months after stroke onset, and proportion of patients who continued taking statins drugs at 12 months after stroke onset. | 12 months after stroke onset
  Medication persistence at 12 months. Persistence at 12 months is defined as continuing a therapy or class of therapy at 12 months follow-up. Subjects prescribed an individual medication at discharge but who were not taking that medication at follow up were defined as "nonpersistent". Persistence for the specified medication classes (antiplatelet, statins) was defined in the same way; however, subjects were considered persistent if there was a switch to another medication within the same class.
Proportion of patients who continued taking antiplatelet drugs in 1 year after stroke onset, and proportion of patients who continued taking statins drugs in 1 year after stroke onset. | 1 year after stroke onset
  Patients who took statins and antiplatelet medications at 3, 6 and 12 months follow-up were regarded as persistent during one year after stroke onset.
Recurrence of ischemic stroke in three months after stroke onset | 3 months after stroke onset
  Recurrence of IS was defined as a new focal neurological deficit of vascular origin lasting >24 hours and without hemorrhage on computed tomography or MRI of the brain.
Recurrence of ischemic stroke in six months after stroke onset | 6 months after stroke onset
  Recurrence of IS was defined as a new focal neurological deficit of vascular origin lasting >24 hours and without hemorrhage on computed tomography or MRI of the brain.
Recurrence of ischemic stroke in 12 months after stroke onset | 12 months after stroke onset
  Recurrence of IS was defined as a new focal neurological deficit of vascular origin lasting >24 hours and without hemorrhage on computed tomography or MRI of the brain.

SECONDARY OUTCOMES:
clinical prognosis | 3,6,12 months
  Death(including Vascular death and non-vascular death); Nonfatal myocardial infarction; Nonfatal hemorrhagic stroke; Severe disabilities(modified Rankin Scale≥4)

CONTACTS AND LOCATIONS:
Overall Officials: yongjun wang, MD, Principal Investigator — Beijing Tian Tan Hospital, Capital Medical University, Beijing, China
Locations (1):
- Beijing Tian Tan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Crocker TF, Brown L, Lam N, Wray F, Knapp P, Forster A. Information provision for stroke survivors and their carers. Cochrane Database Syst Rev. 2021 Nov 23;11(11):CD001919. doi: 10.1002/14651858.CD001919.pub4. PMID 34813082